CLINICAL TRIAL: NCT04280653
Title: An Open-Label, Multi-Center, Clinical Study Evaluating the Effect of the NDE L68 StableFit® Punctal Plug on the Tear Lake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDE68-19-01
Record Dates: First submitted 2020-01-31; First posted 2020-02-21 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NDE L68 StableFit® punctal plug (Experimental): Each study subject that qualifies at the baseline visit will receive an NDE L68 StableFit® punctal plug in the lower punctum in one of their eyes. All study plugs will remain in the study subject's lower punctum for a period of 28 + 4 days after insertion
  Interventions: Device: NDE L68 StableFit® Punctal Plug

INTERVENTIONS:
Device: NDE L68 StableFit® Punctal Plug — Tear lake evaluation of the planned study eye, prior to insertion of the Punctal Plug and then tear lake evaluation at days 7 and 28 after punctal plug insertion.
  Other Names: L-shaped Punctal Plug

SUMMARY:
To evaluate the effect of the NDE L68 StableFit® punctal plug on the tear lake.

DETAILED DESCRIPTION:
This is a Non-Significant Risk (NSR) medical device, multi-center, open-label clinical study. Each study subject that qualifies at the baseline visit will receive an NDE L68 StableFit® punctal plug in the lower punctum in one of their eyes. All study plugs will remain in the study subject's lower punctum for a period of 28 + 4 days after insertion.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female subject, 18 years of age or older, in good general health at the time of the baseline examination, who may or may not have a mild to moderate dry eye condition
2. A subject must be able to read, comprehend and be willing to give HIPAA authorization and informed consent
3. A subject must be willing to have a punctal plug inserted in the lower punctum of one of their eyes
4. A subject must be willing to comply with all study instructions, agree to make all office appointments, and complete the entire course of the study

Exclusion Criteria:

1. A subject with a history of complications, adverse events, trauma or disease in the nasolacrimal area, whether or not it was due to punctal plug wear, including but not limited to dacryocystitis, inflammation or canaliculitis in the planned study eye
2. A subject with a history of intolerance to punctal plugs
3. A subject with structural lid abnormalities (e.g., ectropion, entropion) in the planned study eye
4. A subject with any clinically significant lid, conjunctival or corneal findings in the planned study eye at the baseline visit
5. A subject with a severe dry eye condition
6. A subject experiencing epiphora in the planned study eye
7. A subject experiencing any clinically significant ocular pain or discomfort in or around either eye at the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Eye Institute-Edgewood, Edgewood, Kentucky
  - Ophthalmic Consultants of Long Island, Garden City, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal healthy volunteers were interviewed to determine if they were interested in participating in the study. Recruitment was in the ophthalmologist office by the study staff.
Pre-assignment Details: There was no wash out or run-in period in this study. There was only 1 arm in this study.
Period: Overall Study
Arm/Group | NDE L68 StableFit® Punctal Plug
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NDE L68 StableFit® Punctal Plug
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  20-<25 years | 1
  25- <30 years | 4
  30-<35 years | 4
  45- <50 years | 2
  55- <60 years | 2
  60- <65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Investigators' Evaluation of the Tear Lake; Comparison of Baseline Result to 7 Days
Description: The primary study endpoint will be the comparison of the tear lake volume at baseline with the tear lake volume at each follow-up visit. The tear lake will be evaluated using a slit lamp micrometer, the micrometer will be oriented vertically and centered on the lower lid margin at the middle of the lower lid. The tear lake will be measured using the slit lamp micrometer from the lid margin to the superior border of the lower tear lake and measured to 0.1 mm.
  The average mean percent change from baseline tear lake volume was compared to that at 7 days.
Time Frame: 7 days
Measure: Mean (Full Range); unit: mean percent change from baseline
Arm/Group | NDE L68 StableFit® Punctal Plug
Number analyzed (Participants) | 15
mean percent change from baseline | 129 [125 to 166]

2. Primary Outcome: Investigators' Evaluation of the Tear Lake; Comparison of Baseline Result to 28 Days
Description: The primary study endpoint will be the comparison of the tear lake volume at baseline with the tear lake volume at each follow-up visit. The tear lake will be evaluated using a slit lamp micrometer, the micrometer will be oriented vertically and centered on the lower lid margin at the middle of the lower lid. The tear lake will be measured using the slit lamp micrometer from the lid margin to the superior border of the lower tear lake and measured to 0.1 mm.
  The average mean percent change from baseline tear lake volume was compared to that at 28 days.
Time Frame: 28 days
Measure: Mean (Full Range); unit: mean percent change from baseline
Arm/Group | NDE L68 StableFit® Punctal Plug
Number analyzed (Participants) | 15
mean percent change from baseline | 143 [113 to 166]

3. Secondary Outcome: Investigator's Evaluation \ of the Subject's Acceptance of the NDE L68 StableFit® Punctal Plug, Comparison of Baseline Result to 28 Days
Description: Questionnaire
Time Frame: 28 days
Population: The subjects were interviewed at the final visit (28 days) by the Investigator and rated the acceptability of the punctal plug as Very acceptable/Acceptable/somewhat Acceptable/Unacceptable/extremely unaccable
Measure: Count of Participants; unit: Participants
Arm/Group | NDE L68 StableFit® Punctal Plug
Number analyzed (Participants) | 15
Participants
  Very Acceptable | 7
  Acceptable | 7
  Somewhat Acceptable | 1
  Somewhat Unacceptable | 0
  Unacceptable | 0
  Extremely Unacceptable | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the period of the study, 28 days.
Description: To assess subject's qualifications for enrollment and safety of the punctal plug, the investigator evaluated:
  1. Visit 1 Record any clinically significant Ocular Pain or Discomfort Record any clinically significant slit-lamp findings (lid, conjunctival, corneal) At the conclusion of the baseline visit, did the subject experience an adverse device event (ADE)
  2. Follow-up Visits Record any clinically significant slit-lamp findings (lid, conjunctival, corneal) Record ADE since last visit
Arm/Group | NDE L68 StableFit® Punctal Plug
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NDE L68 StableFit® Punctal Plug (N=15)
Clinically significant slit-lamp findings (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After final publication or not published within 12 months following the conclusion of the last of the multi-center sites, and only with written consent of, and review and comment by, the Sponsor, any publication/lecture manuscripts proposed by the Study Center or the Investigator which are to make public any findings, data or results of the Study or any ancillary study must be submitted to the Sponsor for its review, and comment at least ninety days prior to submission for publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT04280653/Prot_SAP_000.pdf